CLINICAL TRIAL: NCT03052400
Title: Efficacy of Mifepristone in Males With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: End of Funding
Sponsor: Charles Drew University of Medicine and Science (Other)
Responsible Party: Principal Investigator, Stanley Hsia, Associate Professor of Medicine, Charles Drew University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-04-2482
Record Dates: First submitted 2017-02-08; First posted 2017-02-14 (Actual); Results first posted 2022-10-19 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes Mellitus; Insulin Resistance
Keywords: type 2 diabetes mellitus; insulin resistance; mifepristone; glucocorticoids
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mifepristone 600 mg daily (Experimental): Mifepristone 300 mg po daily x 2 weeks, followed by mifepristone 600 mg po daily x 10 weeks
  Interventions: Drug: Mifepristone 600 mg daily
- Placebo (Placebo Comparator): Matching, blinded placebo 1 tablet po daily x 2 weeks, followed by matching, blinded placebo 2 tablets po daily x 10 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mifepristone 600 mg daily — Glucocorticoid receptor antagonist
  Other Names: Korlym
  Arms: Mifepristone 600 mg daily
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
Randomized, double blind, placebo-controlled clinical trial examining the efficacy and safety of mifepristone 600 mg daily in male subjects with type 2 diabetes mellitus, not associated with Cushing's syndrome

DETAILED DESCRIPTION:
Randomized, double blind, placebo-controlled clinical trial examining the efficacy and safety of mifepristone 600 mg daily in male subjects with type 2 diabetes mellitus, not associated with Cushing's syndrome, and sub-optimally controlled on basal insulin, with or without prandial insulin and/or maximally-tolerated doses of metformin.

ELIGIBILITY:
Inclusion criteria:

* Males
* Age 18-65 inclusive
* Established T2DM for ≥ 1 year
* Taking stable doses (≤ 20% change in total daily insulin dose within 2 months prior to screening) of basal insulin, with or without prandial insulin (total daily dose must be ≤ 200 units)
* Baseline hemoglobin A1c (HbA1c) 8.0%-10.5%

Exclusion criteria:

* No use of any anti-hyperglycemic agents (oral or injectable) other than metformin or insulin
* No history or clinical suspicion of type 1 diabetes mellitus
* No concurrent chronic use of any corticosteroids by any route and for any indication, or concurrent conditions that may require the initiation of glucocorticoids during the study
* No concurrent lipid-lowering medications whose levels are dependent on CYP3A pathway clearance (e.g., simvastatin, lovastatin, atorvastatin, fluvastatin and rosuvastatin) should either be washed out for at least one month prior to enrollment and/or switched to alternative LDL-cholesterol lowering agents (e.g., pravastatin or ezetimibe) for at least one month.
* No contraindications or known intolerance to mifepristone
* No concurrent use of strong CYP3A inhibitors (e.g., cyclosporine, ergotamine, fentanyl, quinidine, sirolimus, tacrolimus, imidazole antifungals, HIV protease inhibitors, certain macrolide antibiotics)
* No concurrent use of CYP3A inducers (e.g., phenytoin, phenobarbital, carbamazepine, rifampin)
* No concurrent use of medications that may prolong the QT interval (e.g., selected antipsychotics and antidepressants, quinolone antibiotics)
* No daily use of warfarin or non-steroidal anti-inflammatory agents
* Baseline K+ and Mg+2 within the laboratory normal ranges, with or without oral K+ and/or Mg+2 supplementation
* Fasting plasma glucose (FPG) averaging < 280 mg/dL and without polyuria or polydipsia
* No symptomatic hypoglycemia averaging > once per day
* Able and willing to perform self-monitoring of blood glucose (SMBG)
* Mean BP < 140 mmHg systolic or 90 mm Hg diastolic
* Baseline LDL-cholesterol < 200 mg/dL if on lipid-lowering therapy or < 250 mg/dL while not on lipid-lowering therapy
* Fasting triglycerides ≤ 500 mg/dL if on lipid-lowering therapy
* HDL-cholesterol ≥ 25 mg/dL
* No known history of prostate cancer, or elevated level of prostate-specific antigen (PSA) at screening
* Estimated GFR ≥ 30 mL/min
* No concurrent endocrinopathies that have not been stabilized with replacement or other definitive therapies (including known adrenal insufficiency regardless of replacement therapy, cortisol < 5 μg/dL at screening)
* No active hemolytic anemias or hemoglobin variants that render the measurement of HbA1c potentially unreliable
* No other clinically significant hepatic, cardiovascular (including known personal or family history of, or risk factors for long-QT syndrome, QTcF prolongation on ECG > 500 ms), infectious (including HIV or any viral hepatitis), inflammatory, neoplastic or other systemic disease that may contraindicate the change of lipid-lowering therapy, renders mifepristone unsafe, or otherwise confounds data interpretation
* Subjects not likely to start other drugs that may influence the study's outcomes (e.g., weight loss agents)
* Subjects who are able and willing to comply with all components of the study protocol, attend all scheduled follow-up visits, or who do not present other foreseeable barriers that might make the implementation of the protocol problematic or confound data interpretation

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley H Hsia, MD, Principal Investigator — Charles Drew University of Medicine and Science
Locations (1):
- Charles Drew University of Medicine and Science, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing as per NIH funding requirements
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication
Access Criteria: Contact investigator

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mifepristone 600 mg Daily | Placebo
Started | 4 | 4
Completed | 3 | 3
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mifepristone 600 mg Daily | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (6.6) | 55.4 (1.2) | 52.6 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6
Hemoglobin A1c [Mean (Standard Deviation); unit: Percentage of hemoglobin] | 9.8 (0.8) | 9.8 (0.9) | 9.8 (0.8)
Diabetes duration [Mean (Standard Deviation); unit: Years] | 11.7 (8.8) | 14.0 (2.0) | 12.9 (5.8)
Basal insulin daily dose [Mean (Standard Deviation); unit: Units per day] | 73.3 (19.4) | 65.0 (39.5) | 69.2 (28.2)
Body weight [Mean (Standard Deviation); unit: kg] | 107.6 (46.5) | 99.8 (4.5) | 103.7 (29.9)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 39.3 (15.0) | 36.3 (6.6) | 37.8 (10.5)

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c
Description: Glycemic lowering
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: Percentage of hemoglobin
Arm/Group | Mifepristone 600 mg Daily | Placebo
Number analyzed (Participants) | 3 | 3
Percentage of hemoglobin | -2.4 (1.2) | -1.5 (1.4)

2. Secondary Outcome: Weight
Description: Weight in kg
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: kg, change from baseline
Arm/Group | Mifepristone 600 mg Daily | Placebo
Number analyzed (Participants) | 3 | 3
kg, change from baseline | 1.4 (1.4) | 0.5 (3.3)

3. Secondary Outcome: Body Mass Index
Description: Body mass index in kg/m^2
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: kg/m^2, change from baseline
Arm/Group | Mifepristone 600 mg Daily | Placebo
Number analyzed (Participants) | 3 | 3
kg/m^2, change from baseline | 0.6 (0.5) | 0.0 (1.3)

4. Secondary Outcome: Systolic BP
Description: Systolic blood pressure
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: mm Hg, change from baseline
Arm/Group | Mifepristone 600 mg Daily | Placebo
Number analyzed (Participants) | 3 | 3
mm Hg, change from baseline | 3.0 (8.7) | -3.7 (1.2)

5. Secondary Outcome: Diastolic BP
Description: Diastolic blood pressure
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: mm Hg, change from baseline
Arm/Group | Mifepristone 600 mg Daily | Placebo
Number analyzed (Participants) | 3 | 3
mm Hg, change from baseline | -4.3 (8.5) | -3.7 (5.5)

6. Secondary Outcome: LDL-cholesterol
Description: Low-density lipoprotein cholesterol
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: mg/dL, change from baseline
Arm/Group | Mifepristone 600 mg Daily | Placebo
Number analyzed (Participants) | 3 | 3
mg/dL, change from baseline | -1.3 (18.2) | -9.7 (19.3)

7. Secondary Outcome: Cortisol
Description: Serum cortisol level (AM)
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: mg/dL, change from baseline
Arm/Group | Mifepristone 600 mg Daily | Placebo
Number analyzed (Participants) | 3 | 3
mg/dL, change from baseline | 18.8 (9.0) | -0.9 (0.9)

8. Secondary Outcome: ACTH
Description: Serum adrenocorticotrophic hormone level (AM)
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: pg/mL, change from baseline
Arm/Group | Mifepristone 600 mg Daily | Placebo
Number analyzed (Participants) | 3 | 3
pg/mL, change from baseline | 56.0 (39.8) | -8.3 (11.2)

9. Secondary Outcome: Uric Acid
Description: Serum uric acid level
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: mg/dL, change from baseline
Arm/Group | Mifepristone 600 mg Daily | Placebo
Number analyzed (Participants) | 3 | 3
mg/dL, change from baseline | -0.8 (0.6) | 1.1 (0.4)

10. Secondary Outcome: PSA
Description: Prostate-specific antigen level
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: ng/mL, change from baseline
Arm/Group | Mifepristone 600 mg Daily | Placebo
Number analyzed (Participants) | 3 | 3
ng/mL, change from baseline | -0.3 (0.2) | 0.1 (0.2)

11. Secondary Outcome: Hypoglycemic Events
Description: Symptomatic mild and severe hypoglycemic events
Time Frame: Baseline to 3 months
Measure: Number; unit: number of events
Arm/Group | Mifepristone 600 mg Daily | Placebo
Number analyzed (Participants) | 3 | 3
number of events | 22 | 31

12. Secondary Outcome: Adverse Events
Description: Non-hypoglycemia-related adverse events
Time Frame: Baseline to 3 months
Measure: Number; unit: number of events
Arm/Group | Mifepristone 600 mg Daily | Placebo
Number analyzed (Participants) | 3 | 3
number of events | 6 | 2

13. Secondary Outcome: Basal Insulin Dose
Description: Total daily basal insulin dosage
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: Units of insulin per day
Arm/Group | Mifepristone 600 mg Daily | Placebo
Number analyzed (Participants) | 3 | 3
Units of insulin per day | -1.3 (16.0) | 0.7 (17.9)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse events not including hypoglycemia
Arm/Group | Mifepristone 600 mg Daily | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone 600 mg Daily (N=3) | Placebo (N=3)
Worsening of heart failure (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone 600 mg Daily (N=3) | Placebo (N=3)
Work-related injury (Social circumstances) | 1 (1) | 2 (2)
Myalgias (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Prolonged QT Interval (Cardiac disorders) | 1 (1) | 0 (0)
Peripheral edema (Cardiac disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Administrative barriers and pandemic closures limited enrollment, curtailed several secondary outcome measures, and caused early termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT03052400/Prot_SAP_000.pdf